CLINICAL TRIAL: NCT02748759
Title: Early Mobilization of Knee Joint After ACL Reconstructive Surgery Comparing Continuous Passive Motion Versus Manual Passive Mobilization
Brief Title: Early Mobilization of Knee Joint After ACL Surgery. Continuous Passive Motion Versus Manual Passive Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jesús Montesinos Muñoz (Other)
Collaborators: Fundació Eurecat (Other)
Responsible Party: Sponsor-Investigator, Jesús Montesinos Muñoz, Medical Doctor, Althaia Xarxa Assistencial Universitària de Manresa
Organization: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CEIC 13/106
Record Dates: First submitted 2016-04-15; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Continous Passive Motion; Manual Physical Therapy; Range of Motion, Articular; Anterior Cruciate Ligament Reconstruction; Rehabilitation; Kaltenborn Manual Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EXP 1: Manual mobilization / CPM (Active Comparator): Patients were subjected to a manual mobilization using the Kaltenborn approach, in which 15 tibiofemoral glides were applied by a physiotherapist. After a pause of 5 minutes, the patient was collocated in a commercially available CPM device (Kinetec Advanced Prima) and received 15 repetitions of flexo-extension.
  Interventions: Device: CPM; Other: Manual mobilization
- EXP 2: CPM / Manual mobilization (Active Comparator): Patients were collocated in a commercially available CPM device (Kinetec Advanced Prima) and received 15 repetitions of flexo-extension. After a pause of 5 minutes, patients were subjected to a manual mobilization using the Kaltenborn approach, in which 15 tibiofemoral glides were applied by a physiotherapist.
  Interventions: Device: CPM; Other: Manual mobilization

INTERVENTIONS:
Device: CPM — 15 repetitions of flexo-extensión with a commercially available CPM device (Kinetec Advanced Prima)
Other: Manual mobilization — Manual mobilization using the Kaltenborn approach, in which 15 tibiofemoral glides were applied by a physiotherapist

SUMMARY:
Anterior Cruciate Ligament (ACL) injuries by trauma are a prevalent pathology. In the USA, about 200.000 injuries are estimated per year, half of which implicate a total rupture of the ligament. Data indicates that the number of ACL injuries is increasing in young athletes and presents a common problem, especially people playing agility sports.

One of the most widely used methods for the post-surgical mobilization after ACL is the use of Continuous Passive Motion (CPM) devices. These machines are meant to drain residual fluid from the articulation and maintain the mobility of the joint and muscles in the knee. Even though studies show that, an early mobilization after surgery is beneficial to the rehabilitation of the knee joint, recent studies are questioning the efficiency of the CPM when compared with the goal of application. While literature suggests that efficacy of CPM are related with the magnitude of knee flexion and the Range of Motion (ROM) achieved some studies show that the range of motion measured by the CPM is considerably less than the actual ROM.

As other therapy that provides an effective mobilization of the knee joint, the Specific Manual Physical Therapy method (Kaltenborn method) takes in account the physiological combination of rotation and gliding of the two joint surfaces. This technique mobilizes the femorotibial joint by controlling the tibial plateau anteroposterior during flexion and posteroanterior during extension of the knee. Therefore, in the past 30 years there are not studies comparing ROM measurements obtained with CPM and manual physical therapy methods.

It is hypothesized that the benefits of the early passive mobilization after ACL reconstructive surgery are diminished by the limited efficacy of currently used CPM devices. The aim of our study was to determine the range of motion achieved with the passive mobilization using a CPM device compared with a manual method (Kaltenborn method) and to assess that ROM measurements provided by the CPM correlates the real ROM.

ELIGIBILITY:
Inclusion Criteria:

* Rupture of Anterior cruciate ligament
* Ligamentoplasty with partial meniscectomy when necessary using arthroscopy technique

Exclusion Criteria:

* Patients operated after three weeks post-injury because of greater risk of arthrofibrosis
* Patients who had medical complications during surgery
* Patients unable to understand the study protocol and those unwilling to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Knee Range of Motion (ROM) angle | Fifteen hours after surgery
  Maximum knee flexion angle minus the maximum knee extension angle obtained from 15 repetitions of flexo-extension. Measurements were obtained by CPM device and an external goniometer
Knee maximum flexion | Fifteen hours after surgery
  Maximum knee flexion obtained form 15 repetitions of flexo-extensión. Measurements were obtained by CPM device and an external goniometer
Knee maximum extension | Fifteen hours after surgery
  Maximum knee extension obtained form 15 repetitions of flexo-extensión. Measurements were obtained by CPM device and an external goniometer

SECONDARY OUTCOMES:
Pain | Fifteen hours after surgery
  Pain reported by the patient according to Visual Analogic Scale
Fluid volumen drained (ml) | Fifteen hours after surgery
  Fluid volume drained during procedure (ml)
Time (seconds) | Fifteen hours after surgery
  Overall time spent in manual mobilization and CPM mobilization

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Montesinos, MD, Principal Investigator — Althaia Xarxa Assistencial de Manresa
Locations (1):
- Althaia Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided